CLINICAL TRIAL: NCT00593359
Title: The Effect of Lactated Ringer's Solution Versus Albumin and the Alpha-2 Agonist Brimonidine Versus Placebo on Intraocular Pressure During Prone Spine Surgery
Brief Title: Intraocular Pressure During Spine Surgery
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 07-571
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Intraocular Pressure
Keywords: Spinal surgery; Prone spinal surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: Lactated Ringer's replacement for blood loss and placebo eye drops
- B: Lactated Ringer's replacement for blood loss and brimonidine eye drops
- C: Albumin replacement for blood loss and placebo eye drops;
- D: Albumin replacement for blood loss and brimonidine eye drops

SUMMARY:
This study will compare the effect of two intravenous solutions on eye pressure during spine surgery in the following groups:

Group A - Lactated Ringer's replacement for blood loss and placebo eye drops

Group B - Lactated Ringer's replacement for blood loss and brimonidine eye drops

Group C - Albumin replacement for blood loss and placebo eye drops

Group D - Albumin replacement for blood loss and brimonidine eye drops

DETAILED DESCRIPTION:
Patients will be administered either brimonidine eye drops, or placebo eye drops, preoperatively, on the day of surgery and during surgery. Eye pressure will be measured before surgery, every 30 minutes throughout your surgery and every hour for 4 hours following surgery. Subjects will be evaluated before surgery and on days 5, 8, 15 after surgery. During these evaluations, the subject will be asked questions about recovery and his/her eyes will be checked by an ophthalmologist and vision will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Spine surgery with instrumentation in prone position expected to last at least 5 hours;
* Anticipated blood loss ≥ 1L
* Age 18-80 years old;
* ASA physical status I-III.

Exclusion Criteria:

* History of increased intraocular pressure or glaucoma;
* Diabetic retinopathy;
* Heart failure or serious left ventricular dysfunction;
* Abnormal preoperative fundus examination;
* Creatinine > 2 mg/dL;
* Patient refuses blood transfusion or albumin administration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spinal surgery in the prone position for at least 5 hours.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the maximum intraocular pressure at any time during surgery. | 15 days post surgery

SECONDARY OUTCOMES:
Intraocular pressure as a function of surgical duration; Velocity of retrobulbar blood flow; Facial edema and or chemosis; Time to extubation; Duration of recovery Correlation between Dpp and FTc. | 15 days post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States